CLINICAL TRIAL: NCT00004991
Title: Brain Activation During Developmental Speech Production and Speech Perception
Brief Title: Study of Brain Activity During Speech Production and Speech Perception
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000095; 00-N-0095
Record Dates: First submitted 2000-03-18; First posted 2000-03-20 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-08-31

CONDITIONS: Developmental Articulation Disorder; Stuttering
Keywords: Functional Magnetic Resonance Imaging; Stuttering; Speech Perception; Speech Production; Phonology; Development; Motor Control; Neural Networks; Phonological Disorders
MeSH Terms: conditions — Articulation Disorders; Stuttering; Speech Sound Disorder

SUMMARY:
The purpose of this study is to gain a better understanding of the brain's activity and organization in the development of speech disorders. It will compare brain activity in people with normal speech development with those who stutter or who have a phonological disorder (a deficit in how the brain processes speech sounds).

Stuttering and phonological disorders emerge during the critical period of speech development between 2.5 and 12 years of age. During this period, the brain is much more adaptable for speech development than it is after puberty. This study will examine how the brain organization for speech production and perception develops normally during the critical period and how the normal pattern is altered when stuttering and phonological disorders become chronic problems, persisting throughout life.

Volunteer adults and children with and without speech disorders may participate in this study. Eligibility screening will include a brief neurological and physical examination and tests to determine normal speech or a speech disorder. The speech testing will be videotaped. The subject will speak aloud, describe pictures, recall words or numbers, imitate speech sounds and words, and perform some listening tests.

Study participants will undergo magnetic resonance imaging (MRI) to study brain activity. For this procedure, the subject lies on a stretcher that is moved into a donut-shaped machine with a strong magnetic field. During the MRI scan, the subject will perform simple tasks, such as listening to speech or other sounds and saying nonsense words. The procedure should take less than 60 minutes, and usually takes from 20 to 40 minutes.

DETAILED DESCRIPTION:
This is a study of two developmental speech production disorders, which emerge during the critical period of speech development between 2.5 and 12 years of age. During this critical period there is considerably greater brain plasticity for speech functioning which disappears following puberty. Our purpose is to determine how normal brain organization for speech production and perception develops during the critical period and how this normal pattern is altered when stuttering and phonological disorders become chronic problems, persisting throughout the life span. Functional MRI and magnetoencephalography (MEG) are non-invasive methodologies suitable for research in these disorders in children. New methodologies using fMRI and MEG provide the first opportunity for the study of speech production both in normally developing children as well as children and adults with stuttering and/or phonological disorders. Our hypothesis is that, with development, the brain organization for speech production becomes less distributed involving fewer brain regions, and that phonological processing mechanisms become lateralized to the left hemisphere during the critical period of speech development. This research will address whether the brain regions involved in speech are more diffuse and less selective in persons who develop chronic stuttering and phonological disorders, leading to a less efficient dynamic system for speech production.

ELIGIBILITY:
* INCLUSION CRITERIA:

To address the 15 hypotheses formulated for this research, several subject groups will be studied. The functional activation patterns of normal right-handed adults will be compared with normally developing right-handed children and adolescents (ages 6-17) during tasks involving speech segmentation (into phonemes) and speech formulation. All will be native speakers of American English without foreign language use in the home. Corresponding subject groups will be adults and children with stuttering or phonological processing disorders who are right-handed native speakers of American English. Our aim will be to determine how brain function for speech perception and production change during completion of the critical period for speech development and how these systems differ in children with disorders of speech control and phonology who continue to have problems during this period.

EXCLUSION CRITERIA:

A subject will be excluded if he/she has a contraindication to MR scanning such as the following: aneurysm clip; implanted neural stimulator; implanted cardiac pacemaker or autodefibrillator; cochlear implant; ocular implant or foreign body (e.g. metal shavings or splinters); insulin pump; shrapnel, bullet or shot wound; artificial heart valve; tattooed makeup; prostheses of ferromagnetic material; surgical metal clips in the brain, eye or on blood vessels; implanted drug infusion device. The LSS otolaryngologist, Pamela Kearney, M.D., or LSS nurse practitioner Patti Henshel, C.R.N.P., will screen participants with the NMR Center Safety Screening Questionnaire, which also includes additional items such as intraventricular shunts, transdermal medication patches, wire sutures, bone/joint pins, screws, nails, plates, and body piercings. Dr. Kearney or Ms. Henshel will approve or disapprove participation in the study based on her judgement of the MR compatibility of these items, using published guides including Shellock & Kanal (1994) and Shellock (2001). Other exclusion criteria are claustrophobia, pregnancy (as determined by pregnancy testing at NIH's Clinical Center on the day of scanning); aphasia or dysarthria, language and/or cognitive functioning lower than 2 standard deviations below the age-adjusted mean value on screening tests, speech reception thresholds greater than dB; non-native American English speech development; developmental exposure to a language other than English in the home, and medications that affect central nervous system function at time of fMRI scanning. If a potential participant elects to withdraw from medications, this must be done under the care of the participant's own physician prior to participation in this protocol. Medication withdrawal is not part of this study.

Additional exclusion criteria for developmental stuttering only include: language and/or cognitive functioning lower than 1 standard deviation below the age-adjusted mean value on screening tests, left-handedness on the Edinburgh handedness questionnaire; movement disorders (e.g., Huntington disease, chorea, myoclonus, Gilles de la Tourette syndrome, Parkinson's disease, progressive supranuclear palsy, and neuroleptic-induced syndromes), brain tumors, history of traumatic brain injury with loss of consciousness, genetic diseases of the CNS (e.g., chromosomal diseases, metabolic disorders, diffuse sclerosis), chronic infections of the nervous system (e.g., bacterial, vial, parasitic, fungal and yeast), ataxias (inherited and acquired), myopathies (e.g., progressive muscular dystrophies, familial periodic paralysis, congenital disorders of muscle, myoglobinuria, polymyositis), disorders of the neuromuscular junction (e.g., myasthenia gravis), demyelinating diseases (e.g., multiple sclerosis, central pontine myelinolysis), other brain abnormalities, schizophrenia, alcoholism, long-lasting drug dependence, major and/or bipolar depression, obsessive-compulsive disorder, vocal fold paralysis or paresis, joint abnormality, or neoplasm, and history of swallowing disorders, airway obstruction.

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 411
Dates: Start 2000-03-14; Primary Completion 2009-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Wise R, Chollet F, Hadar U, Friston K, Hoffner E, Frackowiak R. Distribution of cortical neural networks involved in word comprehension and word retrieval. Brain. 1991 Aug;114 ( Pt 4):1803-17. doi: 10.1093/brain/114.4.1803. PMID 1884179
- [Background] Klein D, Milner B, Zatorre RJ, Meyer E, Evans AC. The neural substrates underlying word generation: a bilingual functional-imaging study. Proc Natl Acad Sci U S A. 1995 Mar 28;92(7):2899-903. doi: 10.1073/pnas.92.7.2899. PMID 7708745
- [Background] Muller RA, Behen ME, Rothermel RD, Muzik O, Chakraborty PK, Chugani HT. Brain organization for language in children, adolescents, and adults with left hemisphere lesion: a PET study. Prog Neuropsychopharmacol Biol Psychiatry. 1999 May;23(4):657-68. doi: 10.1016/s0278-5846(99)00024-x. PMID 10390724